CLINICAL TRIAL: NCT07240818
Title: Tissue Sample Comparison Between 22G FNB Needle and a New EUS Core Needle Biopsy Device for Pancreatic Lesions: A Single Center Prospective Randomized Pilot Trial
Brief Title: Comparison of FNB to EUS-CNB for Pancreatic Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2321881
Record Dates: First submitted 2025-09-11; First posted 2025-11-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diagnosis of a Pancreaticobiliary Disorder; Biopsy; EUS Guided Biopsy
Keywords: FNB; EUS-CNB; Endodrill; EUS guided biopsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study participant (patient) and pathologist reviewing the biopsy specimen will be masked. The endoscopist performing the procedure will not be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EUS-FNB (Active Comparator): This arm will undergo biopsy via the standard of care, which involves EUS-guided biopsy using the 22-gauge FNB needles
  Interventions: Procedure: EUS-FNB
- EUS-CNB (Experimental): This arm will undergo biopsy with the novel EUS-CNB device
  Interventions: Device: endoscopic ultrasound guided biopsy with core needle biopsy device

INTERVENTIONS:
Device: endoscopic ultrasound guided biopsy with core needle biopsy device — The EUS-CBD (Endodrill, Bibb Medical, Lund Sweden) differs from currently available needles (FNB) in that it obtains tissue by drilling into target lesions rather than puncturing them.
  Arms: EUS-CNB
Procedure: EUS-FNB — Biopsy obtain via EUS-FNB
  Arms: EUS-FNB

SUMMARY:
The primary aim of this study is to compare the tissue specimen quality and diagnostic accuracy of biopsies obtained with one puncture of a regular 22 FNB G needle and the motorized EUS CNB device of pancreatic lesions. The secondary aims are to compare the rate of blood contamination in the specimens obtained from biopsies of pancreatic lesions and the overall procedure duration. The hypothesis of this study is that the proportion of cases in which a single puncture of the lesion in question delivers adequate diagnostic tissue is higher with the motorized EUS CNB than with the 22 G FNB.

DETAILED DESCRIPTION:
This study is planned as a single-blind, parallel-group randomized pilot clinical trial (RCT). After receiving informed consent, the eligible subjects will be randomly assigned to two parallel arms. The first arm will be assigned to the 22 FNB G needle with dry suction technique. The second arm will be assigned to the EUS CNB. 15 patients will be assigned to each group. Patients will be prospectively enrolled until the target sample size has been reached.

Patients will be enrolled in a prospective manner at the University of California Davis Medical Center Endoscopy unit. The day of the procedure, the endoscopist performing the procedure will explain the EUS-guided biopsy procedure and the risks of the procedure it as usual. After that, the endoscopist will explain the study, and will acquire informed consent from the patients. The patients will be asked to sign the consent only after the study has been explained and all questions have been answered by the performing physician. The Endoscopist will randomize the study subjects using a random number list generated by a simple block randomization scheme via SAS software by the study statistician, to one of the 2 arms: FNB or EUS CNB. The randomization number will be kept in a sealed opaque envelope in numerical sequence and will also contain a card that specifies which device was used. Following randomization, each patient will be assigned a code corresponding to one of the two arms. This code will be noted and placed in a master spreadsheet that only the study coordinator and/or assigned research personnel will handle.

All the procedures will be performed by a single experienced interventional endoscopist (Antonio Mendoza-Ladd, M.D.) The FNB needle to be used in this trial is a 22-gauge SharkCore™ (MEDTRONIC) FNB needle. The EUS CNB device used for the other arm is the Endodrill © as described above. The procedures will be performed under deep monitored or general anesthesia under the care of an anesthesiologist. Once the lesion is evaluated and located by EUS, the endoscopist will select the shortest pathway, while avoiding blood vessels, to reach the lesion. Under real-time visualization, each lesion will be punctured with a single pass using either the Sharkcore FNB or the Endodrill. A cytotechnologist will then perform a Rapid On-Site Examination (ROSE) evaluation of the tissue fragment obtained with this single pass to determine if tissue is adequate for pathological analysis. Once this is the case, the specimens will be submitted to the pathology lab where a GI pathologist will determine all the tissue-related outcomes using only the first-pass tissue specimen of both devices. The cellularity and blood contamination of the specimen will be assigned according to scales previously described by Gerke et al (9) and Wee et al (I&). A score of 2::2 and 2::4 will be considered adequate for cytological and histological diagnosis, respectively. The pathologists evaluating the sample will be blinded to the type of device used to obtain the specimen.

If the tissue sample is deemed suboptimal in this initial pass, the endoscopist will be allowed to break the protocol and use a different needle and/or technique according to his preference and perform as many passes as needed until ROSE reports diagnostic tissue. All the specimens obtained outside of the study protocol will be analyzed for diagnostic purposes but not for research purposes. Regardless of the number of passes, once the tissue is deemed to be adequate for diagnosis, the procedure will stop.

Data Collection: Multiple measures will be taken (storage of study data in an encrypted file in the UCD DOM server behind the secured network firewall, separate key file from data collection sheet access) to ensure the risk to patient confidentiality is minimized. Patient medical data via chart review of the electronic medical records will only be accessed and reviewed by the 2 primary investigators of this study: Antonio Homero Mendoza Ladd, M.D. and Michael Ladna, M.D. The first round of Data collection will occur during the informed consent process and will include demographic data (age, biological sex, ethnicity, weight, and BMI) and relevant medications (antiplatelet and anticoagulants). The second round of data collection will occur during the procedure and will include lesion location, size, lesion characteristics, perioperative complications/adverse events, procedure duration, number of needle passes, and technical success of the procedure. The third round of data collection will occur during the Rapid On-Site Examination (ROSE) using a tissue fragment obtained via a single needle pass. The remainder of the tissue will be placed in a jar with formalin and will be closed and adequately labeled as a "study specimen". The fourth round of data collection will occur once the final histopathologic interpretation and read of the specimen is completed by the pathologist.

Adverse event monitoring: The patients will be monitored during and shortly after the procedure for adverse events. All the study patients will then be seen in the interventional gastroenterology clinic with the primary endoscopist Dr. Mendoza Ladd (who carried out all the procedures) 1-2 months after the procedure to monitor for adverse events. At this clinic appointment the electronic medical records of the study patient will be reviewed by the primary endoscopist Dr. Mendoza Ladd, and co-investigator Dr. Ladna to assess for adverse events. An independent safety reviewer will also be appointed to monitor adverse events and determine whether they were related or unrelated to the study. Dr. Urayama will be appointed as the independent safety reviewer. All adverse events will be documented and reported immediately to the IRB in accordance with the institutional guidelines.

Withdrawal of subjects: Participants will be informed of their right to withdraw from the study at any time during the informed consent discussion with the patient. In cases where safety concerns arise, the investigator has the authority to remove a participant from the study to protect their health and well-being. Concerns which would warrant involuntary withdrawal of the patient from the study include but are not limited to:

1. hemodynamic instability (defined as hypotension with SBP below 90 or MAP below 65)
2. clinical signs of active infection (fever with temp above 38.0 C, sepsis)
3. acute encephalopathy preventing informed consent
4. clinical signs of acute stroke (new focal neurologic deficits, severe headache, visual deficits)
5. acute hypoxic respiratory failure (defined as hypoxia with spO2 <92% and/or increased supplemental oxygen need from baseline for patients on continuous home O2 supplementation and/or need for emergent intubation and mechanical ventitation)
6. intractable nausea/vomiting not responding to anti-emetic medication administration
7. Patients who did not hold systemic anticoagulation (warfarin, apixaban, dabigatran, rivaroxaban, edoxaban, enoxaparin, fondaparinux) 72 hours before the procedure

ELIGIBILITY:
Inclusion Criteria:

1. Patients who require EUS and tissue sampling of pancreatic solid lesions (size> 2.5 cm)
2. Patients who can give consent

Exclusion Criteria:

1. patients without pancreatic lesions
2. Pregnant females
3. Hematologic and Coagulation disorders (platelets < 50,000/mm3, INR > 2, ANC <1000)
4. Patients with acute pancreatitis in the immediate 2 weeks before the procedure (if the lesion to be biopsied is in the pancreas)
5. Cardiorespiratory dysfunction that precludes sedation
6. patients unable to provide informed consent
7. Previous chemotherapy or radiotherapy for a pancreatic neoplasm
8. Patients who are not candidates for emergency surgery in case complications arise from the biopsy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic specimen | during study intervention
  The percentage of cases achieving an adequate diagnostic yield (defined as a cellularity score of ≥2) after a single needle pass with either the EndoDrill or the 22-G FNB device

SECONDARY OUTCOMES:
Blood contamination of the specimen | during study intervention
  Blood contamination of the biopsy specimen obtained from the first needle pass with either the EndoDrill or 22-G FNB, assessed using the following scoring system, in which higher numerical scores correspond to a lower degree of blood contamination and, consequently, superior biopsy specimen quality:
  0: Only blood
  1. Blood contamination in more than 50% of the slide
  2. Blood contamination from 25 to 50% of the slide
  3. Blood contamination in less than 25% of the slide
cellularity score | during study intervention
  Cellularity score of the biopsy specimen obtained from the first needle pass with either the EndoDrill or 22-G FNB, based on the following grading scale, in which higher numerical scores indicate superior biopsy specimen quality:
  0: Insufficient material. The sample is inadequate for interpretation.
  1. Limited cytologic interpretation. There is some material, but it is insufficient for a reliable diagnosis.
  2. Adequate cytologic interpretation. Sufficient cellular material is available for a basic cytologic diagnosis.
  3. Limited histologic assessment. Allows for a limited evaluation of tissue architecture.
  4. Adequate histologic interpretation. The sample contains sufficient tissue to evaluate the lesion's histology. The total tissue length may be within a single microscopic field.
  5. Excellent histologic interpretation. The sample contains a substantial amount of tissue core, exceeding the length of a single microscopic field.
Procedure Duration | during study intervention
  duration in minutes of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mendoza Ladd A, Alsamman A, Meiklejohn K, Viramontes O. Initial experience with transmural use of a new endoscopic ultrasound electric core needle biopsy device: Case series. Endosc Int Open. 2024 Oct 28;12(10):E1237-E1241. doi: 10.1055/a-2427-2311. eCollection 2024 Oct. PMID 39474489
- [Result] Ding S, Lu A, Chen X, Xu B, Wu N, Edoo MIA, Zheng S, Li Q. Diagnostic accuracy of endoscopic ultrasound-guided fine-needle aspiration: A single-center analysis. Int J Med Sci. 2020 Oct 16;17(17):2861-2868. doi: 10.7150/ijms.48882. eCollection 2020. PMID 33162814
- [Result] Wong T, Pattarapuntakul T, Netinatsunton N, Ovartlarnporn B, Sottisuporn J, Chamroonkul N, Sripongpun P, Jandee S, Kaewdech A, Attasaranya S, Piratvisuth T. Diagnostic performance of endoscopic ultrasound-guided tissue acquisition by EUS-FNA versus EUS-FNB for solid pancreatic mass without ROSE: a retrospective study. World J Surg Oncol. 2022 Jun 24;20(1):215. doi: 10.1186/s12957-022-02682-3. PMID 35751053
- [Result] Swahn F, Glavas R, Hultin L, Wickbom M. The advent of the first electric driven EUS-guided 17 gauge core needle biopsy - A pilot study on subepithelial lesions. Scand J Gastroenterol. 2024 Jul;59(7):852-858. doi: 10.1080/00365521.2024.2336611. Epub 2024 Apr 15. PMID 38618997
- [Result] Gerke H, Rizk MK, Vanderheyden AD, Jensen CS. Randomized study comparing endoscopic ultrasound-guided Trucut biopsy and fine needle aspiration with high suction. Cytopathology. 2010 Feb;21(1):44-51. doi: 10.1111/j.1365-2303.2009.00656.x. Epub 2009 May 18. PMID 19456845